CLINICAL TRIAL: NCT07078669
Title: Comparison of Patient Outcomes With Dyed vs. Undyed Polyglactin Sutures in Cutaneous Surgery
Brief Title: Dyed vs. Undyed Polyglactin Sutures in Cutaneous Surgery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Sarah Campbell, Assistant Professor, West Virginia University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2504138740
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Wound Closure; Suture Materials

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dyed Sutures (Active Comparator): Polyglactin 910 (Vicryl) is an absorbable suture commonly utilized for cutaneous surgery; it is available in both dyed (violet) and undyed forms. This arm designates the Dyed Sutures.
  Interventions: Device: Polyglactin 910 (Dyed)
- Undyed Sutures (Active Comparator): Polyglactin 910 (Vicryl) is an absorbable suture commonly utilized for cutaneous surgery; it is available in both dyed (violet) and undyed forms. This arm designates the Undyed Sutures.
  Interventions: Device: Polyglactin 910 (Undyed)

INTERVENTIONS:
Device: Polyglactin 910 (Dyed) — Half the wound for each participant will be sutured using Polyglactin 910 suture dyed (violet) with colorants such as D&C Violet No. 2 present.
  Arms: Dyed Sutures
Device: Polyglactin 910 (Undyed) — Half the wound for each participant will be sutured using Polyglactin 910 suture Undyed
  Arms: Undyed Sutures

SUMMARY:
Purpose - This exploratory, split-wound study aims to evaluate the potential difference in skin reactions to two different types of sutures, dyed and undyed, used to close wounds after surgery. The study will assess whether dyed sutures to elicit increased tissue reactivity like redness, itching, and scarring and whether undyed sutures may be more optimal for wound healing and cosmetic response. Enrollment into the study and data collection is expected to take approximately 3-6 months. Follow-up visits will be chosen at 2 weeks, 4 weeks, and 3 months post-surgery, which is standard practice for monitoring healing and checking for complications such as infection or abnormal scarring.

Primary Objective - The primary objective is to assess the response of wounds closed with both dyed and undyed sutures after cutaneous surgery to determine if there is a difference in wound healing and tissue reactivity with one compared to the other.

Enrollment into the study and data collection is expected to take approximately 3-6 months. Follow-up visits will be chosen at 2 weeks, 4 weeks, and 3 months post-surgery, which is standard practice for monitoring healing and checking for complications such as infection or abnormal scarring.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a standard of care surgical excision

Exclusion Criteria:

* Patients who are unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Erythema Assessment scale | 2 weeks post-procedure
  Erythema will be assessed on both sides of the surgical wound using a 0-4 Clinical Erythema Assessment scale: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe with 0 being the better outcome and 4 the worst.
Clinical Erythema Assessment scale | 4 weeks post-procedure
  Erythema will be assessed on both sides of the surgical wound using a 0-4 Clinical Erythema Assessment scale: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe with 0 being the better outcome and 4 the worst.
Clinical Erythema Assessment scale | 3 months post-procedure
  Erythema will be assessed on both sides of the surgical wound using a 0-4 Clinical Erythema Assessment scale: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe with 0 being the better outcome and 4 the worst.
Presence of Hypertrophic Scarring | 2 weeks post-procedure
  Percentage of the presence of hypertrophic scarring. Visual clinical assessment of each side of the wound will document the presence or absence of hypertrophic scarring (yes/no). A lower percentage of presence of hypertrophic scarring is better than higher.
Presence of Hypertrophic Scarring | 4 weeks post-procedure
  Percentage of the presence of hypertrophic scarring. Visual clinical assessment of each side of the wound will document the presence or absence of hypertrophic scarring (yes/no). A lower percentage of presence of hypertrophic scarring is better than higher.
Presence of Hypertrophic Scarring | 3 months post-procedure
  Percentage of the presence of hypertrophic scarring. Visual clinical assessment of each side of the wound will document the presence or absence of hypertrophic scarring (yes/no). A lower percentage of presence of hypertrophic scarring is better than higher.
Presence of Suture Extrusion | 2 weeks post-procedure
  Presence of Suture Extrusion: Wound evaluation will record whether sutures are visibly extruding from the skin (yes/no) on each side of the wound, to compare extrusion frequency (percentage of suture extrusion being present) between suture types.
Presence of Suture Extrusion | 4 weeks post-procedure
  Presence of Suture Extrusion: Wound evaluation will record whether sutures are visibly extruding from the skin (yes/no) on each side of the wound, to compare extrusion frequency (percentage of suture extrusion being present) between suture types.
Presence of Suture Extrusion | 3 Months post-procedure
  Presence of Suture Extrusion: Wound evaluation will record whether sutures are visibly extruding from the skin (yes/no) on each side of the wound, to compare extrusion frequency (percentage of suture extrusion being present) between suture types.
Presence of Surgical Site Infection | 2 weeks post-procedure
  Presence of Surgical Site Infection: Wound will be evaluated for signs of infection (e.g. erythema, exudate, tenderness) and recorded as yes/no to compare infection frequency (percentage of infection being present) between suture types.
Presence of Surgical Site Infection | 4 weeks post-procedure
  Presence of Surgical Site Infection: Wound will be evaluated for signs of infection (e.g. erythema, exudate, tenderness) and recorded as yes/no to compare infection frequency (percentage of infection being present) between suture types.
Presence of Surgical Site Infection | 3 Months post-procedure
  Presence of Surgical Site Infection: Wound will be evaluated for signs of infection (e.g. erythema, exudate, tenderness) and recorded as yes/no to compare infection frequency (percentage of infection being present) between suture types.
Presence of Edema | 2 weeks post-procedure
  Presence of Edema: Wound will be evaluated for signs of edema and recorded as yes/no to compare frequency of presence between suture types.
Presence of Edema | 4 weeks post-procedure
  Presence of Edema: Wound will be evaluated for signs of edema and recorded as yes/no to compare frequency of presence between suture types.
Presence of Edema | 3 months post-procedure
  Presence of Edema: Wound will be evaluated for signs of edema and recorded as yes/no to compare frequency of presence between suture types.
Presence of Wound Induration | 2 weeks post-procedure
  Presence of Wound Induration: Wound will be evaluated for signs of edema and recorded as yes/no to compare frequency of presence between suture types.
Presence of Wound Induration | 4 weeks post-procedure
  Presence of Wound Induration: Wound will be evaluated for signs of edema and recorded as yes/no to compare frequency of presence between suture types.
Presence of Wound Induration | 3 months post-procedure
  Presence of Wound Induration: Wound will be evaluated for signs of edema and recorded as yes/no to compare frequency of presence between suture types.
Presence of Hyperpigmentation | 2 weeks post-procedure
  Presence of Hyperpigmentation: Visual observation will determine whether increased pigmentation is present at the wound site and recorded as yes/no to compare frequency of presence between suture types.
Presence of Hyperpigmentation | 4 weeks post-procedure
  Presence of Hyperpigmentation: Visual observation will determine whether increased pigmentation is present at the wound site and recorded as yes/no to compare frequency of presence between suture types.
Presence of Hyperpigmentation | 3 months post-procedure
  Presence of Hyperpigmentation: Visual observation will determine whether increased pigmentation is present at the wound site and recorded as yes/no to compare frequency of presence between suture types.
Presence of Exudate | 2 weeks post-procedure
  Presence of Exudate: Each side of the wound (dyed and undyed) will be checked for exudate (fluid drainage) and recorded as yes/no to assess differences in wound response.
Presence of Exudate | 4 weeks post-procedure
  Presence of Exudate: Each side of the wound (dyed and undyed) will be checked for exudate (fluid drainage) and recorded as yes/no to assess differences in wound response.
Presence of Exudate | 3 months post-procedure
  Presence of Exudate: Each side of the wound (dyed and undyed) will be checked for exudate (fluid drainage) and recorded as yes/no to assess differences in wound response.
Presence of Dehiscence | 2 weeks post-procedure
  Presence of Dehiscence: Each side of the wound (dyed and undyed) will be checked for dehiscence (any separation or opening) at the site of closure and recorded as yes/no to compare frequency of presence between suture types.
Presence of Dehiscence | 4 weeks post-procedure
  Presence of Dehiscence: Each side of the wound (dyed and undyed) will be checked for dehiscence (any separation or opening) at the site of closure and recorded as yes/no to compare frequency of presence between suture types.
Presence of Dehiscence | 3 months post-procedure
  Presence of Dehiscence: Each side of the wound (dyed and undyed) will be checked for dehiscence (any separation or opening) at the site of closure and recorded as yes/no to compare frequency of presence between suture types.
Failure to Epithelialize | 2 weeks post-procedure
  Failure to Epithelialize: Each side of the wound (dyed and undyed) will be evaluated for failure to epithelialize (incomplete skin coverage) and recorded as yes/no to compare differences between suture types.
Failure to Epithelialize | 4 weeks post-procedure
  Failure to Epithelialize: Each side of the wound (dyed and undyed) will be evaluated for failure to epithelialize (incomplete skin coverage) and recorded as yes/no to compare differences between suture types.
Failure to Epithelialize | 3 months post-procedure
  Failure to Epithelialize: Each side of the wound (dyed and undyed) will be evaluated for failure to epithelialize (incomplete skin coverage) and recorded as yes/no to compare differences between suture types.
Presence of Suture Granuloma | 2 weeks post-procedure
  Presence of Suture Granuloma: Granuloma formation at the suture site will be visually identified and recorded as yes/no. Comparison will be made between dyed and undyed sides.
Presence of Suture Granuloma | 4 weeks post-procedure
  Presence of Suture Granuloma: Granuloma formation at the suture site will be visually identified and recorded as yes/no. Comparison will be made between dyed and undyed sides.
Presence of Suture Granuloma | 3 months post-procedure
  Presence of Suture Granuloma: Granuloma formation at the suture site will be visually identified and recorded as yes/no. Comparison will be made between dyed and undyed sides.
Presence of Contact Dermatitis | 2 weeks post-procedure
  Presence of Contact Dermatitis: Contact dermatitis will be assessed and graded on a standardized International Contact Dermatitis Research Group (ICDRG) grading scale: - (none), + (weak), ++ (strong), +++ (extreme), IR (irritant) with none being the best outcome. The grading will be used to compare reactions between the two suture types.
Presence of Contact Dermatitis | 4 weeks post-procedure
  Presence of Contact Dermatitis: Contact dermatitis will be assessed and graded on a standardized International Contact Dermatitis Research Group (ICDRG) grading scale: - (none), + (weak), ++ (strong), +++ (extreme), IR (irritant) with none being the best outcome. The grading will be used to compare reactions between the two suture types.
Presence of Contact Dermatitis | 3 months post-procedure
  Presence of Contact Dermatitis: Contact dermatitis will be assessed and graded on a standardized International Contact Dermatitis Research Group (ICDRG) grading scale: - (none), + (weak), ++ (strong), +++ (extreme), IR (irritant) with none being the best outcome. The grading will be used to compare reactions between the two suture types.
Patient-Rated Pruritus | 2 weeks post-procedure
  Patient-Rated Pruritus: Patient will rate itch severity on each side of the wound using a 0-3 scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe with 0=none being the better outcome.
Patient-Rated Pruritus | 4 weeks post-procedure
  Patient-Rated Pruritus: Patient will rate itch severity on each side of the wound using a 0-3 scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe with 0=none being the better outcome.
Patient-Rated Pruritus | 3 months post-procedure
  Patient-Rated Pruritus: Patient will rate itch severity on each side of the wound using a 0-3 scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe with 0=none being the better outcome.
Patient-Rated Pain/Tenderness | 2 weeks post-procedure
  Patient-Rated Pruritus: Patients will rate pain/tenderness on each side of the wound using a 0-3 scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe with 0=none being the better outcome.
Patient-Rated Pain/Tenderness | 4 weeks post-procedure
  Patient-Rated Pruritus: Patients will rate pain/tenderness on each side of the wound using a 0-3 scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe with 0=none being the better outcome.
Patient-Rated Pain/Tenderness | 3 months post-procedure
  Patient-Rated Pruritus: Patients will rate pain/tenderness on each side of the wound using a 0-3 scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe with 0=none being the better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Camplbell, MD, Principal Investigator — West Virginia University-Dermatology
Locations (1):
- WVU Medicine Waynesburg Dermatology, Waynesburg, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No